CLINICAL TRIAL: NCT04486014
Title: A Comparative Study of the Analgesic Effect of Ultrasound-guided Erector Spinae Plane Block Versus Serratus Anterior Plane Block for Thoracoscopic Sympathectomy Surgeries
Brief Title: Analgesic Effect of Erector Spinae Versus Serratus Anterior Plane Block for Thoracoscopic Sympathectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD.20.04.307
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-09

CONDITIONS: Thoracic Sympathectomy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind (participant) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae plane block (ESP) (Experimental): Patients would receive erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- Serratus anterior plane block (SAP) (Experimental): Patients would receive serratus anterior plane block
  Interventions: Procedure: Serratus anterior plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — Erector Spinae Group (Group E) will receive bilateral ultrasound-guided erector spinae plane block using 30 ml hyperbaric bupivacaine 0.25% will be injected between erector spinae muscle and transverse process of T4
  Arms: Erector spinae plane block (ESP)
Procedure: Serratus anterior plane block — Serratus anterior Group (Group S) will undergo bilateral ultrasound-guided serratus anterior plane block with 30 ml hyperbaric bupivacaine 0.25% will be injected above or below serratus anterior muscle at the level of 4th and 5th rib on the midaxillary line
  Arms: Serratus anterior plane block (SAP)

SUMMARY:
* Thoracic incisions are painful and associated with chronic post-surgical pain and inadequate analgesia is associated with poorer postoperative outcomes. Recent progress has been made in the field of thoracic anesthesia by improving analgesic modalities such as PECS 1 and PECS 2, intercostal plane block, paravertebral regional anesthesia, ultrasound-guided erector spinae and serratus anterior plane block.
* Administered of the local anesthetic in erector spinae plane block is in the interfascial plane between the transverse process of the vertebra and the erector spinae muscles, spreading to multiple paravertebral spaces. It affects both the ventral and dorsal rami and leading to blockage of both visceral and somatic pain.
* Ultrasound-guided serratus anterior plane block is a facial plane block that provides analgesia by blocking of lateral branches of intercostal nerves above or below the serratus plane muscle.
* We hypothesize that the ultrasound-guided erector spinae plane block may have better quality than the serratus anterior plane block for patients undergoing thoracoscopic sympathectomy as erector spinea plane blocks visceral and somatic pain.

DETAILED DESCRIPTION:
Primary palmar hyperhidrosis (PPH) refers to the excessive secretion of exocrine glands on the palms, which is often accompanied by the head, face, or plantar hyperhidrosis. PPH demonstrates no obvious organic cause; however, some patients may feel distressed because their palms sweat more than normal, and such a situation may lead to severe psychological, social, and occupational dysfunction.

Endoscopic thoracic sympathectomy abolishes eccrine sweating in all areas supplied by the postganglionic fibers with its complications which include post-sympathetic neuralgia which is the most important, wound infection, hemorrhage, pneumothorax, horner syndrome, no response to the operation and compensatory hyperhidrosis in non-denervated areas.

Forero described ultrasound-guided erector spinae plane block for treatment of thoracic neuropathic pain and explained it as a peri-paravertebral regional anesthesia technique that has been used for prevention of postoperative pain in various surgeries.

Ultrasound-guided serratus anterior plane block is a facial plane block which provides analgesia by blocking of lateral branches of intercostal nerves above or below the serratus plane muscle. There are few cases and studies in the literature reporting successful analgesia provided by serratus anterior plane block

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists grade I or II physical status

Exclusion Criteria:

* Patients who had coagulopathies
* local infections
* neuropathies
* neuromuscular disease
* psychiatric disease
* history of thoracic surgery
* history of allergy to local anesthetics.
* receiving chronic analgesic therapy
* drug abusers

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
The total analgesic consumption | 1st 24 hours after surgery
  cumulative consumption of opioids during the first postoperative day

SECONDARY OUTCOMES:
Postoperative severity of the pain | every 2 hours for 12hours and then at 16, 20 and 24 hours postoperatively
  Visual analogue scale (0-100),where 0 point is equal to no pain and 100 indicate the worst possible pain
The total amount of fentanyl consumption | 1st 24 hours after surgery
  cumulative consumption of fentanyl during the first postoperative day
The total amount of paracetamol consumption | 1st 24 hours after surgery
  cumulative consumption of paracetamol during the first post operative day
Duration of analgesia | within 24 hours after surgery
  from the end of block till the time for the first analgesic requirement (ketorolac)
Nausea | 1st 24 hours after surgery
  number of patients with nausea
Vomiting | 1st 24 hours after surgery
  number of patients with vomiting
Patient Satisfaction | After 12 and 24 hours after surgery
  evaluated as 5:excellent, 4:very good, 3:good, 2: fair, 1:poor
Heart rate | Intraoperative (every 10 minutes till the end of surgery)
  changes in heart rate
Peripheral oxygen saturation | Intraoperative (every 10 minutes till the end of surgery)
  changes in Peripheral oxygen saturation as measured with pulse oximetry
End-tidal carbon dioxide tension | Intraoperative (every 10 minutes till the end of surgery)
  changes in end-tidal carbon dioxide tension as measured with capnography
systolic blood pressure | Intraoperative (every 10 minutes till the end of surgery)
  changes in systolic blood pressure
diastolic blood pressures | Intraoperative (every 10 minutes till the end of surgery)
  changes in diastolic blood pressure
mean blood pressures | Intraoperative (every 10 minutes till the end of surgery)
  changes in mean arterial blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y Makharita, MD, Study Chair — Professor of Anesthesia and Surgical Intensive care,P; Doaa G Diab, MD, Study Director — Associate Professor of Anesthesia and Surgical Intensive care,
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the study and being accepted for publication.
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients